CLINICAL TRIAL: NCT06884865
Title: A Phase 2, Two-Part, Randomized, Double-Blind, Active-Controlled Study to Assess the Safety and Tolerability of Enekinragene Inzadenovec (PCRX-201) in Subjects With Painful Osteoarthritis of the Knee
Brief Title: A Study to Assess Safety and Tolerability of PCRX-201 in Subjects With Painful Osteoarthritis of the Knee
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201-C-201
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: gene therapy; Knee Pain Arthritis; Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: In Part A (manufacturing process 1), subjects are randomized in a 1:1:1 ratio to Dose A , Dose B , or placebo, each with a predose IA steroid of methylprednisolone acetate.
  In Part B (manufacturing process 2), subjects are randomized in a 1:1:1 ratio to Dose A, Dose B, or placebo, each with a pre-dose IA steroid of methylprednisolone acetate.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part A Dose A (Experimental): Single Intra-Articular injection
  Interventions: Biological: Enekinragene Inzadenovec (PCRX-201)
- Part A, Placebo (Placebo Comparator): Single Intra-Articular injection
  Interventions: Biological: Placebo
- Part B Dose A (Experimental): Single Intra-Articular injection
  Interventions: Biological: Enekinragene Inzadenovec (PCRX-201)
- Part B Dose B (Experimental): Single Intra-Articular injection
  Interventions: Biological: Enekinragene Inzadenovec (PCRX-201)
- Part B Placebo (Placebo Comparator): Part B Placebo
  Interventions: Biological: Placebo
- Part A, Dose B (Experimental): Single Intra-Articular injection
  Interventions: Biological: Enekinragene Inzadenovec (PCRX-201)

INTERVENTIONS:
Biological: Enekinragene Inzadenovec (PCRX-201) — Enekinragene Inzadenovec (PCRX-201) injection
  Arms: Part A Dose A; Part A, Dose B; Part B Dose A; Part B Dose B
Biological: Placebo — Placebo injection
  Arms: Part A, Placebo; Part B Placebo

SUMMARY:
The goal of this clinical trial is to learn if a single knee injection of different doses (Dose A and Dose B) of an investigation product PCRX-201, following steroid pretreatment, is safe and tolerable in male of female patients 45 to 80 years old with osteoarthritis of the knee. It will also learn how the body reacts to the PCRX-201 injection and how effective the treatment is.

Researchers will compare Dose A and Dose B of PCRX-201 versus placebo from Week 1 through Week 52 to assess adverse events. Researchers will also explore how PCRX-201 may impact knee pain and joint function over time.

Participants will be asked to

* Visit the clinic for pretreatment and drug administration
* Visit the clinic for checkups and tests:

  1. Screening through Week 52: intially weekly, bi-weekly, later monthly
  2. Week 53 through Week 260 (Year 5): 8 visits throughout the period

DETAILED DESCRIPTION:
The study will consist of two parts, Part A and Part B, which will use PCRX-201 from two different manufacturing processes. A total of 135 eligible subjects, with painful OA of the index knee will be enrolled. Subjects will be randomly assigned to a treatment dose group, stratified by Kellgren-Lawrence (K-L) Grade, in both parts of the study. Enrollment of subjects with K-L Grade 4 will be capped at 4 subjects per dose group in Part A and 8 subjects per dose group in Part B.

Enrollment of subjects with K-L Grade 2 or 3 will include a minimum of 4 subjects per Grade per dose group in Part A and a minimum of 8 subjects per Grade per dose group in Part B. This study does not require an equal number of subjects between K-L Grade 2 and 3. All eligible subjects will be pretreated with the same dose of methylprednisolone acetate (40 mg) on Day 1 immediately before treatment with PCRX-201 or placebo.

Part A will enroll approximately 45 subjects into 3 dose groups (15 subjects in each treatment group, stratified by K-L Grade as noted above).

Part B will enroll approximately 90 subjects into 3 groups (30 subjects in each treatment group, stratified by K-L Grade as noted above). Enrollment in Part B is dependent upon the availability of study drug developed with manufacturing process 2.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to comply with the study procedures and visit schedule and able to follow verbal and written instructions.
* Subjects must be male or female and 45 to 80 years old, inclusive, at Screening.
* Subjects must exhibit symptoms associated with osteoarthritis of the index knee for ≥12 months before Screening (subject self-reporting is acceptable).
* Subjects must have index knee pain for >15 days over the last month before Screening (subject self-reporting is acceptable).
* Subjects must have failed 2 or more therapies: Restricted physical activity as per Osteoarthritis Research Society International (OARSI) core level recommendation, ie, "structured land-based exercise" (this may include physical therapy), and failure of an additional type of conservative therapy for OA of the index knee, eg, nonselective NSAIDs or COX-2 inhibitors, in the past 12 months.
* Subjects must have a body mass index (BMI) ≤40 kg/m2 at Screening.
* Subjects must have an index knee examination indicating the index knee and the intended injection site area are free of any signs of local or joint infection at Baseline.
* Subjects must have an index knee Average Daily Knee Pain (NRS) between ≥5.0 and ≤9.0 at Screening and Baseline.
* Sexually active subjects of child-bearing potential (SOCBP) and their partners must agree to use effective birth control while in the study
* Subjects must have active synovitis in the index knee as determined by ultrasound Doppler.
* Subjects must exhibit American College of Rheumatology Criteria (clinical and radiological) for osteoarthritis as follows:

  1. Knee pain
  2. At least 1 of the following:

  i. Age >50 years ii. Morning stiffness <30 minutes iii. Crepitus on knee motion c. Osteophytes
* Subjects must have K-L Grade 2, 3, or 4 in the index knee based on X-rays performed during Screening and confirmed by trained radiographers at a central facility before enrollment
* Subjects need to show the presence of moderate or severe synovitis based on 11-point synovitis score using contrast-enhanced MRI

Exclusion Criteria:

* Subjects have any current or prior diagnosis of autoimmune connective tissue disorders, secondary OA conditions, benign synovial tumors, gout/pseudogout, reactive arthritis, RA, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease.
* Subjects have any active systemic or local infection, including infection of the index knee
* Subjects are unable to undergo MRI with contrast MRI
* Subjects with X-ray or MRI exclusionary events
* Subjects have an unstable index knee joint (eg, torn anterior cruciate ligament) within 12 months of Screening
* Subjects have used any approved or investigational IA drug/biologic in index knee within 6 months of Screening (eg, hyaluronic acid, platelet rich plasma, stem cells, prolotherapy, and amniotic fluid injection)
* Subjects are receiving or have received any gene therapy treatment (eg, IL-1Ra) in the past 3 years
* Subjects have used IA steroids ≤3 months before screening

Other protocol-defined criteria apply

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2032-03 (Estimated)

PRIMARY OUTCOMES:
Incidence (number and percent) of treatment-emergent adverse events (TEAEs) for PCRX-201 Dose A and Dose B versus placebo from Week 1 through Week 52 | Week 1 through Week 52.
Incidence (number and percent) of adverse events of special interest (AESIs) for PCRX-201 Dose A and Dose B versus placebo from Week 1 through Week 52 | Week 1 through Week 52.
Incidence (number and percent) of serious adverse events (SAEs) for PCRX-201 Dose A and Dose B versus placebo from Week 1 through Week 52 | Week 1 through Week 52.

SECONDARY OUTCOMES:
Real-time quantitative polymerase chain reaction (qPCR) measurement profile in plasma of PCRX-201 Dose A and Dose B from postdose through Week 8 | Days 1, 4, Weeks 2, 4, 8
Real-time qPCR measurement profile of skin swab samples from Baseline through Week 4. | Days 1, 4, Weeks 2, 4
Assessment of the levels of neutralizing antibodies (NAbs), high-sensitivity C-reactive protein (hs-CRP), and biomarkers of inflammation (eg, interleukin [IL]- 1, cytokines [tumor necrosis factor alpha (TNFα), IL-1β, IL-6, IL-10], and chemokines [IL-8]) | Days 1, 4, Weeks 2, 3, 4,12, 16, 24, 38
Absolute change from baseline in Average Daily Knee Pain (Numerical Rating Scale [NRS]) for PCRX-201 Dose A and Dose B versus placebo. | Weeks 38 and 52
Absolute change from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Score for PCRX-201 Dose A and Dose B versus placebo. | Weeks 38 and 52
Absolute change from baseline in WOMAC Stiffness Score for PCRX-201 Dose A and Dose B versus placebo. | Weeks 38 and 52
Absolute change from baseline in WOMAC Physical Function Score for PCRX-201 Dose A and Dose B versus placebo. | Weeks 38 and 52
Absolute change from Baseline on the Knee Injury and Osteoarthritis Outcome Score (KOOS) function/daily living score for PCRX-201 Dose A and Dose B versus placebo at Weeks 38 and 52. | Weeks 38 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Nino Joy, MD, Study Director — Pacira Pharmaceuticals, Inc
Locations (17):
- United States (17):
  - Osteoporosis Medical Center, Beverly Hills, California
  - Beach Physicians Medical Group Inc., Huntington Beach, California
  - Horizon Clinical Research, La Mesa, California
  - Alliance Clinical West Hills (Focus Clinical Research), West Hills, California
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Journey Research Inc., Oldsmar, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Injury Care Research, LLC, Boise, Idaho
  - Physicians Research Collaboration, Lincoln, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - NY Scientific, Brooklyn, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clinical Trials of South Carolina - Charleston, Charleston, South Carolina
  - Clinical Trials of South Carolina - Columbia, Columbia, South Carolina
  - Zenos Clinical Research, Dallas, Texas
  - Epic Clinical Research, Lewisville, Texas

IPD SHARING:
Plan to Share IPD: Undecided